CLINICAL TRIAL: NCT01759355
Title: Hybrid PET/MR in the Therapy of Cervical Cancer: A Pilot Study
Brief Title: Hybrid PET/MR in the Therapy of Cervical Cancer
Status: Completed | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: LCCC1221
Record Dates: First submitted 2012-12-17; First posted 2013-01-03 (Estimated); Last update posted 2021-12-03 (Actual); Status verified 2021-12

CONDITIONS: Cervix Carcinoma; Cervical Squamous Cell Carcinoma; Cervical Adenosquamous Carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Surgery: Participants undergoing surgical intervention will receive a PET/MR scan prior and following surgery for a total of two (2) scans.
  Interventions: Procedure: FDG PET/MR
- Chemoradiation: Participants undergoing chemoradiation intervention will receive a PET/MR scan prior, during, and following chemoradiation for a total of three (3) scans.
  Interventions: Procedure: FDG PET/MR

INTERVENTIONS:
Procedure: FDG PET/MR — Participants will undergo a FDG, gadolinium enhanced PET/MR scan.
  Other Names: FDG Positron Emission Tomography/Magnetic Resonance Scan

SUMMARY:
This is a two arm, single center feasibility study of 20 patients with non-metastatic cervical cancer managed with surgery and/or chemoradiation therapy at UNC Hospitals. Subjects will undergo PET/MRI scans before, during (chemoradiation group only), and after treatment.

DETAILED DESCRIPTION:
The primary purpose of this study is to evaluate the feasibility of obtaining complete and interpretable hybrid PET/MR images for patients diagnosed with cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Biopsy-proven, previously untreated squamous cell carcinoma, adenosquamous carcinoma, or adenocarcinoma of the uterine cervix
* Clinically visible lesion at least FIGO stage Ib or AJCC 7th edition T1b
* Scheduled to undergo standard of care PET/CT for baseline assessment of disease
* Anticipated to be eligible for curative intent therapy (surgery of chemoradiation therapy) as determined by the patient's primary oncologist
* If female of child-bearing potential, negative serum or urine pregnancy test ≤ 7 dats prior to first PET/MRI
* Informed consent reviewed and signed

Exclusion Criteria:

* History of sever reaction to contrast-enhanced CT scan
* Inability to tolerate MRI (e.g., inability to lie flat > 1 hour)
* Presence of pacemaker, intracranial aneurysm clip, bladder stimulator, cochlear implant or metal near eyes
* Poorly controlled diabetes mellitus
* Creatinine > 1.4 mg/dL or GFR < 30 mL/min
* Body Mass Index (BMI) > 35
* Active vaginal bleeding requiring packing and emergent radiation therapy
* Pregnant or lactating female
* History of a prior malignancy within past 5 years, unless disease free for ≥ 3 years
* Substance abuse, medical, psychological, or social conditions that may interfere with study participation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: UNC Hospitals
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2020-05-28 (Actual); Study Completion 2020-05-28 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who successfully complete PET/MR scans at all study time-points | 2-3 months post-treatment

SECONDARY OUTCOMES:
Sensitivity of PET/MR for baseline disease assessment | pre-treatment
  Estimated proportion of subjects with disease (positive pathology or PET/CT) that have positive PET/MR scans.
Specificity of hybrid PET/MR for baseline disease assessment | pre-treatment
  Proportion of subjects without disease (negative pathology or PET/CT) that have negative PET/MR scans.
Accuracy of hybrid PET/MR for baseline disease assessment | pre-treatment
  Proportion of correct assessments among total population
Detection of disease with PET/MR at each time point | pre-treatment to 2-3 months post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Oldan, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina-Chapel Hill, Chapel Hill, North Carolina, United States